CLINICAL TRIAL: NCT04634968
Title: The Effectiveness of a Brief Motivational Interviewing (MI) Communication Via Instant Massaging on the Reduction of Drug Abuse Among Adolescents in Hong Kong: a Pilot Randomized Controlled Trial
Brief Title: Peer-delivered Follow-up Text Communication After a Brief Motivational Interviewing (MI) for Adolescent Drug Abusers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MedPAC-Pilot
Record Dates: First submitted 2020-11-09; First posted 2020-11-18 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2021-10

CONDITIONS: Drug Abuse; Adolescent Behavior
Keywords: drug abuse; brief motivational interview; peer counselling; instant messaging; adolescent
MeSH Terms: conditions — Substance-Related Disorders; Adolescent Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The interactive Brief MI-based text message communication via instant messaging apps (e.g., WhatsApp, WeChat) will be applied in the intervention group. The chatting function of WhatsApp and WeChat will be used as the intervention platform. The intervention will start on the first day after the participants join the follow-up group. The whole interactive text-communication intervention lasts for 1 month. The frequency of message communication will be at least twice a week. After completing the intervention, participants will be invited to complete an individualized telephone-based interview for collecting further information on the intervention content.
  Interventions: Behavioral: Brief Motivational Interviewing interaction
- control group (Placebo Comparator): The participants in the control group will receive general health communication twice every week via SMS. The communication lasts for 1 month. After completing the intervention, participants will be invited to complete an individualized telephone-based interview for collecting further information on the intervention content.
  Interventions: Behavioral: General health communication

INTERVENTIONS:
Behavioral: Brief Motivational Interviewing interaction — Telephone peer counselling+ Brief Motivational Interviewing interaction, and telephone-based interview after receiving all information.
  Arms: intervention group
Behavioral: General health communication — Telephone peer counselling+ General health communication, and telephone-based interview, and telephone-based interview after receiving all information.
  Arms: control group

SUMMARY:
A pilot randomized control trial will be conducted attaching to the MedPAC services to evaluate the feasibility and acceptability of a Motivational Interviewing (BMI) interaction via instant messaging apps on reducing the drug abuse among youth in Hong Kong.

DETAILED DESCRIPTION:
Youth who persistently abuse substances often experience an array of problems, including academic difficulties, health-related problems (including mental health), poor peer relationships, and involvement with the juvenile justice system. Additionally, there are consequences for family members, the community, and the entire society. Although many youths engage in risky, experimental drug use without developing later life addiction, the early age of first drug use is strongly associated with risk for developing a substance use disorder later in life.

According to the Central Registry of Drug Abuse Sixty-seventh Report in 2018, the total number of reported drug abusers in Hong Kong has been decreasing in last decade, however, about 40% of them were aged 25 or below. Reported by 2017/18 Survey of Drug Use among Students, the number of students claiming to have used drugs has gone up by 23 per cent compared to the last survey. Combining with the two reports, there were lifetime drug-taking 17800 students, while only 471 drug-users aged under 21 were reported. In addition, the 2017 figures revealed that 58% of the abusers took drugs at home/friend's home only, which had increased substantially from 43% in 2008. The statistics above alarm that the drug abuse and the hidden nature of drug-taking among the youth aged 25 or below which cannot be overlooked or undervalued.

The psychological and social factors associated with the initiation and continuation of drug abuse are different for the youth and adult. Previous research has confirmed that the recovery from drug abuse is influenced by the users' intention to change, which is determined directly by their perceptions of anti-drug and their perceived self-efficacy to change. While, drug-abusers' attitude, social influences, and demographic characteristics have more indirect effects on recovery from drug abuse.

Most of the youth drug-abusers reported that the major reasons to take drugs for the first time are "curiosity" and "to seek excitement", which indicated an insufficient anti-drug awareness among the high-risk population. While except for the conform bringing by drug-abusing, social and psychological factors, such as peer identification, depression, anxiety, stress was reported as major reasons for youth to continue using drugs. It prompts us individualized interventions that clearly communicated information about the risks of drug abuse should be designed for the youth.

Government has organized several drug abuse treatment and rehabilitation programme. However, as shown in the report, about 88% of youth drug-abusers had never sought others' help. Except for the feeling that drug giving, absence of problem lead to that they mostly did not consider themselves addicted, which was the major reason for the youth having no awareness to seek for others' help. In addition, consideration about the stigma, fear of not knowing what to expect from the treatment and the whole lifestyle change, and worries about withdrawal symptoms were the main barriers to keep the youth from seeking drug abuse treatment. To bring the usage of drug abuse treatment and rehabilitation programme into full play, these barriers should be resolved for drug-abusing youth.

Considering the reasons above, specifically promoting and supporting service should be developed to increase the anti-drug awareness of the youth, enhancing help-seeking consciousness, and promote treatment and rehabilitation for youth drug-abusers or those exposed to drug abuse.

Telephone counselling is effective in promoting addiction behaviour, both in Hong Kong and overseas. As reported in a previous study, the clients prefer to use online counselling as it was less confronting than traditional forms of counselling by providing a private and emotionally safe environment. Therefore, the telephone format encourages those who are reluctant to get help face-to-face to seek direct anti-drug advice. In addition, the telephone method is proven to be more effective than other health promotion intervention such as mass media as it allows the counsellor to directly interact with the caller, thus addressing the problem at the right moment. Comparing with face-to-face counselling, analyses have consistently reported that telephone counselling allows a large segment of drug-abusers to be reached at a minimal cost. Hence, the use of telephone counselling in helping drug-abusing youth cannot be ignored.

Comparing with general counsellors, there are several advantages using peer as counsellors. There is evidence supporting that the use of peer counsellors can increase the appeal of addiction services to youth users. Since most youths are not eligible to hold positions of power in their society, they find themselves, subject to authority. Such a power differential makes communication between adult and youth difficult. When one is trying to engage the youth in drug abuse prevention initiatives, this power differential manifests itself also as a knowledge gap. The adults' command over jargon and the "science" of drug addiction often acts as a deterrent for the youth who may otherwise willingly engage in debate. Comparing with adults, the equality in power status between the youth makes peer-based risk communication successful. With similar age, peers can address concerns relevant to their experience, which help the high-risk youth to aware of the problem of drug abuse. Explanation and consideration from peers could be more effective in helping drug-abusing youth to eliminate or reduce the fear of unknown to expect from the treatment and the whole lifestyle change, and worries about withdrawal symptoms. Hence, they could be more willing to attempt to seek further help and treatment.

Moreover, a thorough understanding of drug-abusing youth, especially the psychological and social factors that cause them to initiation and continuation of drug abuse, is necessary to design individualized interventions to these drug-abusers. The trained peer counsellors provided individualized advice to the drug-abusing youth to improve their self-efficacy to resist the urge to drug and control over their own behaviour. Peers can better understand the problems that people their age faced such as peer pressure, conflict with parents and teachers and girl-boy relationships. The empathy on the social and psychological problem between the youth could be a good approach for drug-abusing youth to pour out their pressures, which is associated with the prevention of relapse. As stated above, peer counselling could be a potential method in increasing awareness of drug abuse, promoting help-seeking and preventing relapse of drug abuse among the drug-abusing youth.

On the other hand, the collaborator of this project, the Society for the Aid and Rehabilitation of Drug Abusers (SARDA) found in 1961, has rich experience in addiction counselling and drug treatment and rehabilitation. SARDA has seven affiliated treatment and rehabilitation centres and one clinic, which can accept the referral cases who need further treatment and rehabilitation service. The medical doctors in the clinic have sound knowledge of the drug abused, counselling skills, and can handle patients with drug overdose or drug abuse. In addition, medical doctors, experienced counsellors in SARDA will be invited to give lectures in a training programme held for the student counsellors.

ELIGIBILITY:
Inclusion Criteria:

* age 25 years old or below,
* report taking drugs within the past 30 days,
* be able to speak Cantonese, read Traditional Chinese,
* accept to received counseling use messaging apps (such as WhatsApp, WeChat, and SMS text messenger),
* have verbally consented to join the follow-up intervention.

Exclusion Criteria:

* have acute psychosis or other mental problems,
* be undergoing other drug abuse recovery treatment.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-12-04 (Actual)

PRIMARY OUTCOMES:
Changes of drug abuse consumption | 1-month
  The participants' changes of drug abuse consumption between baseline and 1-month follow-up.

SECONDARY OUTCOMES:
Changes of level of readiness to quit | 1-month
  The participants' changes of level of readiness to quit between baseline and 1-month follow-up, measured measured using the Transtheoretical Model of behavior change, including pre-contemplation stage, contemplation stage, decision stage, action stage, and maintenance stage, including pre-contemplation stage, contemplation stage, decision stage, action stage, and maintenance stage.
The rate of changes of level of readiness to quit at 3 month comparing to that at baseline | 3-month
  The participants' changes of level of readiness to quit between baseline and 3-month follow-up, measured using the Transtheoretical Model of Behavior Change, the tool consists of 5 items which include pre-contemplation stage, contemplation stage, decision stage, action stage, and maintenance stage.
The rate of changes of level of readiness to quit at 6 month comparing to that at baseline | 6-month
  The participants' changes of level of readiness to quit between baseline and 6-month follow-up, measured using the Transtheoretical Model of Behavior Change, the tool consists of 5 items which include pre-contemplation stage, contemplation stage, decision stage, action stage, and maintenance stage.
Changes of perceived treatment needs | 1-month
  Participants' changes of the perceived treatment needs between baseline and 1-month follow up measured using the Chinese version of Treatment Needs/Motivation Scales (TCU MOTForm). The The scale consists of 36 items with 5 subscales, namely Problem Recognition (PR), Desire for Help (DH), Treatment Readiness (TR), Pressures for Treatment (PT), and Treatment Needs (TN), which are using a 5-likert score. The score of the scale ranges from 36 to 180, with higher score indicating a higher perceived treatment need.
Changes of perceived treatment needs | 3-month
  Participants' changes of the perceived treatment needs between baseline and 3-month follow up measured using the Chinese version of Treatment Needs/Motivation Scales (TCU MOTForm). The The scale consists of 36 items with 5 subscales, namely Problem Recognition (PR), Desire for Help (DH), Treatment Readiness (TR), Pressures for Treatment (PT), and Treatment Needs (TN), which are using a 5-likert score. The score of the scale ranges from 36 to 180, with higher score indicating a higher perceived treatment need.
Changes of perceived treatment needs | 6-month
  Participants' changes of the perceived treatment needs between baseline and 6-month follow up measured using the Chinese version of Treatment Needs/Motivation Scales (TCU MOTForm). The The scale consists of 36 items with 5 subscales, namely Problem Recognition (PR), Desire for Help (DH), Treatment Readiness (TR), Pressures for Treatment (PT), and Treatment Needs (TN), which are using a 5-likert score. The score of the scale ranges from 36 to 180, with higher score indicating a higher perceived treatment need.
The changes of motivation towards solving the problem | 1-month
  Participants' changes of motivation towards solving the problem between baseline and 1-month follow up measured using the Chinese version of Treatment Needs/Motivation Scales (TCU MOTForm). The The scale consists of 36 items with 5 subscales, namely Problem Recognition (PR), Desire for Help (DH), Treatment Readiness (TR), Pressures for Treatment (PT), and Treatment Needs (TN), which are using a 5-likert score. The score of the scale ranges from 36 to 180, with higher score indicating a higher motivation towards solving the problem.
The changes of motivation towards solving the problem | 3-month
  Participants' changes of motivation towards solving the problem between baseline and 3-month follow up measured using the Chinese version of Treatment Needs/Motivation Scales (TCU MOTForm). The The scale consists of 36 items with 5 subscales, namely Problem Recognition (PR), Desire for Help (DH), Treatment Readiness (TR), Pressures for Treatment (PT), and Treatment Needs (TN), which are using a 5-likert score. The score of the scale ranges from 36 to 180, with higher score indicating a higher motivation towards solving the problem.
The changes of motivation towards solving the problem | 6-month
  Participants' changes of motivation towards solving the problem between baseline and 6-month follow up measured using the Chinese version of Treatment Needs/Motivation Scales (TCU MOTForm). The The scale consists of 36 items with 5 subscales, namely Problem Recognition (PR), Desire for Help (DH), Treatment Readiness (TR), Pressures for Treatment (PT), and Treatment Needs (TN), which are using a 5-likert score. The score of the scale ranges from 36 to 180, with higher score indicating a higher motivation towards solving the problem.
Changes in drug consumption at 3 month comparing to that at baseline | 3-month
  The participants' changes in drug consumption between baseline and 3 months follow-up using using a Structured-Questionnaire gathering the frequency and categoties of drug consumption in the past 30 days. The more frequencies and the more kinds of drug used indicating the higher consumption of drug abuse.
Changes in drug consumption at 6 month comparing to that at baseline | 6-month
  The participants' changes in drug consumption between baseline and 6 months follow-up using using a Structured-Questionnaire gathering the frequency and categoties of drug consumption in the past 30 days. The more frequencies and the more kinds of drug used indicating the higher consumption of drug abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Shuk Ting Cheung, Phd, Study Director — HKU
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient-level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project is completed and the results of the project have been published.
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)

REFERENCES:
- [Result] Saunders B, Wilkinson C, Phillips M. The impact of a brief motivational intervention with opiate users attending a methadone programme. Addiction. 1995 Mar;90(3):415-24. doi: 10.1046/j.1360-0443.1995.90341510.x. PMID 7735025
- [Result] Padwa H, Guerrero EG, Serret V, Rico M, Gelberg L. Adapting substance use brief interventions for adolescents: perspectives of adolescents living with adults in substance use disorder treatment. Subst Abuse Rehabil. 2018 Dec 5;9:137-142. doi: 10.2147/SAR.S177865. eCollection 2018. PMID 30584386
- [Result] de Gee EA, Verdurmen JE, Bransen E, de Jonge JM, Schippers GM. A randomized controlled trial of a brief motivational enhancement for non-treatment-seeking adolescent cannabis users. J Subst Abuse Treat. 2014 Sep;47(3):181-8. doi: 10.1016/j.jsat.2014.05.001. Epub 2014 May 17. PMID 24969735